CLINICAL TRIAL: NCT04065152
Title: Phase II Multicenter Study of Talimogene Laherparepvec in Classic or Endemic Kaposi Sarcoma - KAPVEC
Brief Title: Phase II Multicenter Study of Talimogene Laherparepvec in Classic or Endemic Kaposi Sarcoma
Acronym: KAPVEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P17072019
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Kaposi Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oncolytic immunotherapy (Experimental): Talimogene laherparepvec Dose: 10^6 pfu/ml at week 1 then 10^8/ml at week 4 and every 2 weeks (up to 4ml for each injection) Route: intralesional injection Duration of treatment: 6 months (12 cycles)
  Interventions: Drug: Talimogene laherparepvec

INTERVENTIONS:
Drug: Talimogene laherparepvec — Talimogene laherparepvec

SUMMARY:
Kaposi Sarcoma (KS) is a lymphangioproliferation associated with human herpes virus 8 (HHV8) promoted by immunosuppression. HIV-related KS and iatrogenic posttransplantation KS are treated by immune restoration, in association with local or systemic therapies as chemotherapies if required. Conversely in classic and endemic KS, the underlying relative immunosuppression cannot be directly targeted. Treatment is poorly codified, mostly based on surgery or radiotherapy for localized KS. Most aggressive forms with visceral involvement are treated with chemotherapies or interferon, which give at best 30-60% of transient responses and may not be well tolerated in elderly patients.

Talimogene laherparepvec is the first oncolytic immunotherapy approved by the FDA, in metastatic or unresectable melanoma with injectable nodal or cutaneous lesions. It is designed to induce tumor regression of injected lesions through direct lytic effects, and of uninjected lesions through induction of systemic antitumor immunity.

In Merkel cell carcinoma (MCC), another virus-induced tumor, treatment with PD-1/PD-L1 axis inhibitors have proven efficacy, thus providing a proof of principle that immunotherapy could be effective in virus-induced tumors. Two cases of metastatic MCC successfully treated with talimogene laherparepvec were recently reported, suggesting that talimogene laherparepvec may also be an effective therapeutic option. Considering the high immunogenicity of viral epitopes in KS tumors, the role of the immune evasion in the development of KS, and the cutaneous manifestations (>90% of patients) that can be easily injected, classic and endemic KS is a good tumor model to be targeted with talimogene laherparepvec. The main objective is to assess whether talimogene laherparepvec is clinically inactive (partial+complete response probability π0<10%) or truly active (partial+complete response probability π1>40%) in classic and endemic Kaposi sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Classic or endemic histologically confirmed Kaposi Sarcoma (KS) that is progressive, but does not require a systemic therapy ;
* Injectable and measurable disease, defined as:

  * At least 2 cutaneous lesion ≥10mm in its largest diameter, in a not previously irradiated field;
  * At least 2 other cutaneous lesion ≥10mm in their largest diameter available for repeated cutaneous biopsies, in a not previously irradiated field.
  * Clusters of small lesions with edge to edge distance <2 mm, if the biggest diameter of each cluster meet the 2 previous criteria.
* Be willing to provide tissue from cutaneous biopsy;
* At least 4 weeks washout for all KS specific therapies including topical treatment, chemotherapy, radiotherapy and immunotherapy including interferon;
* Provide written, informed consent prior to the performance of any study specific procedures;
* Be more than 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function:

  * Haematological : Absolute neutrophil count (ANC) ≥1500/mm3; Platelets ≥100 000/mm3; haemoglobin≥ 8 g/dL;
  * Renal: Serum creatinine ≤ 1.5 x upper limit of normal (ULN), OR calculated creatinine clearance ≥ 40mL/min for subject with creatinine levels > 1.5 x ULN.
  * Hepatic: AST (SGOT) and ALT (SGPT) ≤ 2.5xULN, serum total bilirubin ≤ 1.5xULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels >1.5xULN.
  * PT≤1.5; PTT (TCA) ≤1.5
* Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication
* Have a health insurance.

Exclusion Criteria:

* Known history of organ transplantation or HIV (HIV 1/2 antibodies detected at selection);
* Symptomatic visceral involvement of KS including brain metastases;
* Active autoimmune disease that requires systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo, type I diabetes mellitus, hypothyroidism, psoriasis non requiring systemic treatment are permitted to enrol;
* Evidence of clinically significant immunosuppression such as the following: primary immunodeficiency state such as Severe Combined Immunodeficiency Disease; concurrent opportunistic infection;
* Receiving systemic immunosuppressive therapy including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrolment;
* Active herpetic skin lesions or prior complications of HSV-1 infection (eg, herpetic keratitis or encephalitis);
* Intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use;
* Previous treatment with talimogene laherparepvec or any other oncolytic virus;
* Prior radiotherapy in which the fields overlap the injection sites;
* Prior immunosuppressive, chemotherapy, radiotherapy, biological cancer therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to KS therapy administered more than 28 days prior to enrollment.
* Prior therapy with tumor vaccine;
* Received live vaccine within 28 days prior to enrolment;
* Currently treatment with another investigational device or drug study, or less than 28 days since ending treatment with another investigational device or drug study(s);
* Acute or chronic active hepatitis B (HbS Ag detected) or C infection (HCV RNA detected) at inclusion;
* Known additional malignancy that is currently progressing or requires active treatment within the last 3 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer;
* Sensitivity to any of the products or components to be administered ;
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial and 3 months after the last dose of talimogene laherparepvec;
* Subjects who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or infants under the age of 3 months, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec.
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
* Female subject of childbearing potential who are unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec.
* Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Best overall response | 6 months
  Best overall response rate (BORR) defined by the occurrence of complete response or partial response of the injected lesions following PGA criteria (PGA 0 to 4) recorded from the start of treatment until 6 months or the beginning of any other specific therapy for Kaposi sarcoma if it occurs before 6 months.
  PGA score:
  Score and category Description 0: completely clear Complete relief of symptoms; 100% of improvement
  1. almost clear Marked improvement of all clinical symptoms as compared with baseline with residual signs (≥90% and <100%)
  2. marked improvement Significant improvement of symptoms (≥75% and <90%)
  3. moderate improvement Moderate improvement between score 2 and 4.
  4. slight improvement Improvement of signs and symptoms as compared with baseline (<50% and ≥25%) but remaining signs of active KS
  5. no change Clinical signs and symptoms unchanged from baseline (+-25%)
  6. worse Clinical signs and symptoms deteriorated from baseline (≥25% of deterioration)
Overall survival | 6 months
  delay between inclusion and death from any cause
Best overall response M3 | 3 months
  Best overall response rate (BORR) defined by the occurrence of complete response or partial response of the injected lesions following PGA criteria (PGA 0 to 4) recorded from the start of treatment until 6 months or the beginning of any other specific therapy for Kaposi sarcoma if it occurs before 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Dermatologie Hopital Saint-Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided